CLINICAL TRIAL: NCT07044024
Title: An Observational Clinical Study to Evaluate the Efficacy of the CeraVe Skin Care Line in Improving Mild to Severe Acne on the Face
Brief Title: An Observational Clinical Study to Evaluate the Efficacy of the CeraVe Skin Care Line
Status: Not yet recruiting | Type: Observational
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Other Study IDs: C25005055
Record Dates: First submitted 2025-06-15; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide; Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with GEA Class 1: Patients with GEA Classification 1 will be assigned to use CeraVe Blemish Control Cleanser in combination with CeraVe Blemish Control Gel.
  Interventions: Combination Product: CeraVe
- Patients with GEA Class 2: Patients with GEA Classification 2 will be assigned to use CeraVe Blemish Control Cleanser in combination with CeraVe Facial Moisturising Lotion and topical medicine.
  Interventions: Combination Product: CeraVe
- Patients with GEA Class 3: Patients with GEA Classification 3 will be assigned to use CeraVe Foaming Facial Cleanser in combination with CeraVe Facial Moisturising Lotion and topical medicine.
  Interventions: Combination Product: CeraVe
- Patients with GEA Class 4 or above: Patients with a GEA classification of 4 and above will be assigned to use CeraVe Hydrating Facial Cleanser in combination with CeraVe Moisturising Cream in combination with commonly used sunscreen products in combination with oral medications.
  Interventions: Combination Product: CeraVe

INTERVENTIONS:
Combination Product: CeraVe — Patients with GEA classification 1 will be assigned to use CeraVe Blemish Control Cleanser in combination with CeraVe Blemish Control Gel.
  Patients in GEA Class 2 will be assigned to use CeraVe Blemish Control Cleanser in combination with CeraVe Facial Moisturising Lotion in combination with topical medications.
  Patients with GEA classification 3 will be assigned to use CeraVe Foaming Facial Cleanser in combination with CeraVe Facial Moisturising Lotion in combination with topical medications.
  Patients with a GEA classification of 4 and above will be assigned to use CeraVe Hydrating Facial Cleanser in combination with CeraVe Moisturising Cream in conjunction with a commonly used sunscreen product in combination with an oral medication.
  Other Names: Topical acne medications; Oral medications for acne

SUMMARY:
This is an observational clinical study to evaluate the efficacy of the CeraVe Skin Care product line in improving mild to severe facial acne. Primary Objective: To evaluate the efficacy of CeraVe Skincare products in improving mild to severe facial acne through clinical observation by dermatologists of skin conditions before and after the use of the test product kit during the course of acne medication, as well as to collect concurrent feedback on the quality of life of this population and their experience with and satisfaction with the test product. Secondary objectives: 1. To collect feedback on the experience, satisfaction and quality of life improvement of CeraVe products through subjective evaluation of the subjects after using the products, in order to gain a deeper understanding of the comprehensive performance of the products in actual application; 2. To verify the tolerance of CeraVe products through clinical evaluation of the facial skin condition before and after the use of the products by dermatologists; 3. To evaluate the effectiveness of CeraVe products in improving acne. CeraVe is a dermatologist's clinical assessment of facial skin conditions before and after use to verify the tolerability and safety of CeraVe's skin care products. The study is designed to enroll approximately 240 male and female study participants aged 13 years or older with mild to severe facial acne, with a minimum sample size of 200 subjects based on a 15% dropout rate during the trial period and a protocol violation rate of no more than 5%. Participants entering the study will be classified as having mild, moderate, or severe acne according to the Global Evaluation Acne Grading Scale (GEA) (mild-grade 1 or grade 2, moderate-grade 3, severe-grade 4 or higher), with a sample size of mild acne:moderate acne:severe acne of approximately 1:1:1. The study was conducted over an 8-week period with 3 visits. They were conducted at the baseline visit (T0), week 4 follow-up (T4w) and week 8 follow-up (T8w). The window period was ±1 day for the week 4 (T4w) visit and ±2 days for the week 8 (T8w) visit. The primary evaluation parameters included: clinical assessment and product tolerance assessment by the dermatologist, patient self-assessment and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Chinese males and females, age eligible greater than or equal to 13 years old;
* Be in good health and free from any other chronic disease or disease under treatment;
* Be judged by a dermatologist at the Baseline visit:

Mild, moderate, or severe acne according to the Global Evaluation Acne Grading Scale (GEA)11,12 (Mild - Grade 1 or Grade 2) Acne Grading Scale (GEA) - Scale 1 or 2, Moderate - Scale 3, Severe - Scale 4 or above);

* Initiation of acne treatment within the last 3 months with medications that include, but are not limited to, the following

  1. Topical medications: benzoyl peroxide (BPO), retinoic acid, adapalene, isotretinoin, azelaic acid, 0.1% adapalene/BPO. b) Topical medications: benzoyl peroxide (BPO), retinoic acid, adapalene, isotretinoin, azelaic acid, adapalene 0.3% adapalene/BPO, retinoic acid/clindamycin, BPO/clindamycin;
  2. Oral medications: antibiotics, spironolactone, isotretinoin, etc; If Global Evaluation Acne Grading Scale (GEA) classification is ≥2, continuous use of the above medications for at least 2 weeks prior to the baseline visit is required.

     If the Global Evaluation Acne Grading Scale (GEA) is ≥2, acne treatment with the above medications should be continued for at least 2 weeks before the baseline visit; If oral medication is used, acne treatment should be continued for at least 4 weeks prior to the baseline visit.

     Exclusion Criteria:
* Adult female study participants who intend to plan a pregnancy, or who are pregnant, breastfeeding, within 6 months of delivery, or who are unwilling to take the necessary precautions to avoid pregnancy;
* Study participants who are currently enrolled in another clinical study or have been enrolled in another clinical study within 3 months;
* Study participants who have undergone physical, chemical, or cosmetic surgery within 3 months prior to enrollment;
* Systemic diseases with severe organ damage, cardiovascular diseases, liver or kidney dysfunction, malignant tumors, chronic diseases with unstable control, acute infectious diseases, major surgeries or traumas, psychological and psychiatric disorders, or other diseases that require topical or systemic use of medications or treatments that have an effect on acne;
* The study site is associated with other skin disorders (atopic dermatitis, rosacea, rosacea, eczema, etc.) or the presence of other skin conditions that interfere with evaluation (birthmarks, scarring, etc.);
* Participants in the study have a history of allergic contact dermatitis caused by cleansers (facial cleansers)/moisturizers;
* History of allergy or severe allergy to the products (Sensitive Skin products) and related ingredients provided in the study;
* Study participants who are unable to follow compliance requirements, or who are known to be unable to attend visits on time, or who are unwilling to comply with the study protocol arrangements for the duration of the study;
* Any clinical presentation or other illness in the required observation area that, in the opinion of the investigator, may affect the study product assessment or results.
* Study participants had received medical aesthetic treatments (including but not limited to photofacial type treatments, fruit acid resurfacing, etc.) within 3 months prior to enrollment.

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Male or Female Study Participants Aged 13 Years or Older with Mild to Severe Acne on the Face
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-06-27 (Estimated); Primary Completion 2025-09-14 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patients' GEA grading before and after use of the trial product kit | Baseline visit, week 4 visit, week 8 visit
  The Global Evaluation Acne Grading Scale (GEA) is a clinical tool used to assess the severity of acne. The following are the specifics and criteria of the GEA grading scale.
  A score of 0 indicates clean skin with no lesions and possible hyperpigmentation or erythema.
  A score of 1 indicates almost clean skin, almost no lesions, occasionally visible, scattered open or closed pimples, almost no papules. 2 indicates mildly recognizable, almost no papules.
  A score of 2 represents mildly recognizable acne involving no more than half of the face, with a few open or closed pimples, a few papules and pustules.
  A score of 3 represents moderate acne involving more than half of the face, with many open or closed pimples, numerous papules and pustules, and possibly a nodule.
  A score of 4 represents severe acne involving the entire face, with many open or closed pimples, numerous papules and pustules, and occasional nodules.
  A score of 5 represents highly inflammatory acne covering the entire face
The physician evaluates the subject's skin condition by filling out a scale | Baseline visit, week 4 visit, week 8 visit
  The doctor evaluates the subject's skin condition by completing a scale, which is rated on a scale of 0-4 (0=no symptoms, 4=very severe) and includes: sebum secretion, enlarged pores, dryness, flakiness, erythema, itchiness, burning, stinging.
Self-assessment questionnaires on quality of life completed by subjects | Baseline visit, week 4 visit, week 8 visit
  A self-assessment questionnaire of quality of life was completed by the subjects, using a scale of 1-4, (1=not at all, 4=strongly agree), which included whether the subject was bothered by acne, whether acne had an impact on the subject's daily life, socialization, and so on.

SECONDARY OUTCOMES:
The physician assesses the subject's tolerance and satisfaction of the investigational product by completing a scale. | Week 4 visit, week 8 visit
  The physician assesses the subject's tolerance of the investigational product by completing a scale, a 0-4 rating scale (0=not applicable, 4=strongly agree), which includes: whether the subject is a better candidate for the investigational product than for other products; and whether the investigational product is helpful to the patient and whether they were satisfied with the study product.
Questionnaire for patients to assess their own tolerance and satisfaction with the study product | Week 4 visit, week 8 visit
  Patient Assessment of Their Tolerance and Satisfaction with the Study Product Questionnaire, a 0-4 scale questionnaire, (0=not applicable, 4=strongly agree), which included: whether they preferred the study product over other products; whether the study product helped acne, and whether they were satisfied with the study product